CLINICAL TRIAL: NCT02753179
Title: Quality of Life and Dynamic Visual Acuity in Patients With Bilateral Vestibulopathy: the Impact of Covert-saccades
Brief Title: Covert-saccades, Dynamic Visual Acuity and Quality of Life
Acronym: COSQOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 69HCL15_0746
Record Dates: First submitted 2016-04-25; First posted 2016-04-27 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Vestibular Diseases
Keywords: Bilateral vestibular hypofunction; Video Head Impulse Test; Covert-saccades; Quality of life; Dynamic visual acuity
MeSH Terms: conditions — Vestibular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bilateral vestibular hypofunction (Experimental): Patients suffering from chronic bilateral vestibular hypofunction.
  Interventions: Other: Head Impulse Tests; Other: Dynamic visual acuity Test (DVAT); Other: VEMPs & VEMPo; Other: Dizziness Handicap Inventory; Other: Oscillopsia severity questionnaire

INTERVENTIONS:
Other: Head Impulse Tests — Head Impulse Tests are performed by the clinician who holds the patient's head in his hands, while he is looking straight at an earth-fixed target; then by turning the patient's head abruptly and unpredictably to the left or right, up or down through a small angle (only 10-20 degrees - not a large angle). 20 impulses in each directions (6) will be performed.
Other: Dynamic visual acuity Test (DVAT) — Dynamic visual acuity Test (DVAT) assesses visual acuity during head movement relative to baseline static visual acuity. DVA will be assessed actively during self-generated rotations of the head in different directions.
Other: VEMPs & VEMPo — VEMPs & VEMPo are sound evoked muscular contractions of the neck or eye. They are recorded using an evoked response computer, a sound generator, and surface electrodes to pick up neck or eye muscle activation.
Other: Dizziness Handicap Inventory — Dizziness Handicap Inventory is a questionnaire that identify difficulties that patient may be experiencing because of dizziness, yielding to a score ranging from 0 to 100
Other: Oscillopsia severity questionnaire — Oscillopsia severity questionnaire is a 9 items questionnaires that identify oscillopsia in different circumstances.

SUMMARY:
Patients with chronic bilateral vestibular hypofunction may suffer from a visual instability during head movement called oscillopsia. Visual consequence of vestibular deficit can lead to a severe impairment of their quality of life. However, correcting saccades during rapid head movement, called covert-saccades, have been more recently identified. These saccades, which occur during the head movement in patients with vestibular hypofunction, present a very short latency. They could compensate for the lack of vestibular-ocular reflex and greatly decrease oscillopsia and visual impairment. The objective of this study is to evaluate the potential functional benefice of these compensatory movements in a population of 20 patients with chronic bilateral areflexia, in a cross-sectional study.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral Vestibular Hypofunction (BVH) with at least two of the tree following criteria

  * Mean peak slow phase velocity of 5°/s or less in bilateral bithermal (30 and 44°C) caloric irrigations
  * Pathologic Head-impulse test
  * VOR gain of <0.25 on rotatory chair tests
* Disorder present for over 6 month
* Comprehension of the experiments instructions
* Patient consent

Exclusion Criteria:

* Corrected Visual Acuity lower than 5/10
* Other conditions leading to oscillopsia or ataxia
* Oculomotor palsy, ocular instability in primary position
* Cervical rachis pathology with instability
* Cochlear Implants
* Non-stabilized medical disease
* Pregnant women
* Patients under tutelage

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Frequency of covert-saccades | Day 0
  Frequency of covert saccades corresponds to the total amount of covert-saccades divided by the total amount of head impulse tests multiplied by 100.

SECONDARY OUTCOMES:
Quality of life assessed with the Dizziness Handicap Inventory | Day 0
  Dizziness Handicap Inventory is a questionnaire that identify difficulties that patient may be experiencing because of dizziness, yielding to a score ranging from 0 to 100
Dynamic visual acuity | day 0
  Dynamic visual acuity is a measure of threshold for binocular reading of letters that are presented on a screen during head impulse test
Oscillopsia severity questionnaire score | day 0
  Oscillopsia severity questionnaire is a 9 items questionnaires that identify oscillopsia in different circumstances. A mean item score gives an oscillopsia severity score ranging from 1 to 5, yielding to a total score ranging from 0 to 45
Latency of covert-saccades | Day 0
  Latency of covert saccades correspond to the time between the beginning of head impulse and the initiation of the first covert-saccade

CONTACTS AND LOCATIONS:
Overall Officials: Caroline TILIKETE, MD, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Unité de Neuro-Ophtalmologie Hôpital Neurologique, Bron, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hermann R, Pelisson D, Dumas O, Urquizar C, Truy E, Tilikete C. Are Covert Saccade Functionally Relevant in Vestibular Hypofunction? Cerebellum. 2018 Jun;17(3):300-307. doi: 10.1007/s12311-017-0907-0. PMID 29248983